CLINICAL TRIAL: NCT06474299
Title: Dual Use Cessation: A MOST Screening Trial to Identify Effective Interventions to Help People Who Smoke and Vape
Brief Title: The Avenues Study: Dual Use Cessation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0019; R01CA290895 (NIH); A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); Protocol Version 5/13/2025 (Other: UW Madison)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation; Electronic Cigarette Use
Keywords: ENDS; Cessation
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Varenicline; Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: 2x2x2 factorial screening trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Varenicline, Dual Focused, 1 session (Active Comparator)
  Interventions: Drug: Varenicline; Behavioral: Dual Focused Cessation Counseling; Other: Counseling Intensity: 1 Session
- Varenicline, Dual Focused, 4 sessions (Active Comparator)
  Interventions: Drug: Varenicline; Behavioral: Dual Focused Cessation Counseling; Other: Counseling Intensity: 4 Sessions
- Varenicline, Smoking Focused, 1 session (Active Comparator)
  Interventions: Drug: Varenicline; Behavioral: Smoking Focused Cessation Counseling; Other: Counseling Intensity: 1 Session
- Varenicline, Smoking Focused, 4 sessions (Active Comparator)
  Interventions: Drug: Varenicline; Behavioral: Smoking Focused Cessation Counseling; Other: Counseling Intensity: 4 Sessions
- Nicotine Patches, Dual Focused, 1 session (Active Comparator)
  Interventions: Drug: Nicotine patch; Behavioral: Dual Focused Cessation Counseling; Other: Counseling Intensity: 1 Session
- Nicotine Patches, Dual Focused, 4 sessions (Active Comparator)
  Interventions: Drug: Nicotine patch; Behavioral: Dual Focused Cessation Counseling; Other: Counseling Intensity: 4 Sessions
- Nicotine Patches, Smoking Focused, 1 session (Active Comparator)
  Interventions: Drug: Nicotine patch; Behavioral: Smoking Focused Cessation Counseling; Other: Counseling Intensity: 1 Session
- Nicotine Patches, Smoking Focused, 4 sessions (Active Comparator)
  Interventions: Drug: Nicotine patch; Behavioral: Smoking Focused Cessation Counseling; Other: Counseling Intensity: 4 Sessions

INTERVENTIONS:
Drug: Varenicline — 0.5 mg pill once a day for the first 3 days and then increase to a 0.5 mg pill twice a day (at least 8 hours apart) for 4 days prior to the TQD. On the 8th day (the TQD), participants will increase to their target maintenance dose of a 1 mg pill twice daily
  Arms: Varenicline, Dual Focused, 1 session; Varenicline, Dual Focused, 4 sessions; Varenicline, Smoking Focused, 1 session; Varenicline, Smoking Focused, 4 sessions
Drug: Nicotine patch — Following package inserts starting on the TQD, participants who smoke >10 cigarettes per day at baseline will be given 8 weeks of 21 mg nicotine patches, followed by 2 weeks of 14 mg patches, and 2 weeks of 7 mg patches. Participants who smoke ≤10 cigarettes per day at baseline will be given 10 weeks of 14 mg nicotine patches followed by 2 weeks of 7 mg patches.
  Arms: Nicotine Patches, Dual Focused, 1 session; Nicotine Patches, Dual Focused, 4 sessions; Nicotine Patches, Smoking Focused, 1 session; Nicotine Patches, Smoking Focused, 4 sessions
Behavioral: Dual Focused Cessation Counseling — Dual Focused Cessation Counseling will focus on quitting both smoking and vaping. Specifically, participants will be instructed to change smoking and vaping patterns (e.g., not smoking or vaping in specific places such as the car or at specific times of day) prior to quitting and to practice cessation coping strategies (e.g., distraction techniques, getting social support).
  Arms: Nicotine Patches, Dual Focused, 1 session; Nicotine Patches, Dual Focused, 4 sessions; Varenicline, Dual Focused, 1 session; Varenicline, Dual Focused, 4 sessions
Behavioral: Smoking Focused Cessation Counseling — Smoking Focused Cessation Counseling will focus on quitting smoking and using ENDS as a harm reduction strategy (i.e., using ENDS as a substitute for cigarettes).
  Arms: Nicotine Patches, Smoking Focused, 1 session; Nicotine Patches, Smoking Focused, 4 sessions; Varenicline, Smoking Focused, 1 session; Varenicline, Smoking Focused, 4 sessions
Other: Counseling Intensity: 1 Session — Participants assigned to one session will complete a single, 15-20 minute, session at Visit 2 (1 week pre-TQD).
  Arms: Nicotine Patches, Dual Focused, 1 session; Nicotine Patches, Smoking Focused, 1 session; Varenicline, Dual Focused, 1 session; Varenicline, Smoking Focused, 1 session
Other: Counseling Intensity: 4 Sessions — Participants assigned to intensive counseling will have four, 15-20-minute sessions.
  Arms: Nicotine Patches, Dual Focused, 4 sessions; Nicotine Patches, Smoking Focused, 4 sessions; Varenicline, Dual Focused, 4 sessions; Varenicline, Smoking Focused, 4 sessions

SUMMARY:
The overarching goal of this research is to determine the most effective approach for helping dual users of cigarettes and electronic nicotine delivery systems (ENDS) quit smoking. 500 participants will be enrolled and can expect to be on study for 12 months.

DETAILED DESCRIPTION:
To be efficient and maximize translation potential, the investigators will use the efficient Multiphase Optimization Strategy (MOST) to identify an optimal intervention to help people who use both cigarettes and ENDS quit smoking cigarettes. As such, in this randomized 2x2x2 factorial screening trial, the investigators will examine three intervention factors:

1. Pharmacotherapy (varenicline vs. nicotine patch)
2. Counseling Intensity (4 vs. 1 session)
3. Counseling Approach (Dual Focused vs. Smoking Focused).

The Dual Focused counseling approach will encourage participants to quit their ENDS use as part of their smoking cessation attempt. The Smoking Focused counseling approach will encourage participants to quit smoking but not vaping and to use their ENDS strategically to deal with urges in service of harm reduction. There is theoretical and empirical support for these pharmacologic and counseling approaches and intensities.

Participants (N=500) will be dual users of cigarettes (>4 cigs/day for the last 6 months) and ENDS (vape weekly for at least 6 months) who are motivated to quit smoking and willing try to quit vaping, if asked to do so. Participants will be randomized to receive either varenicline or nicotine patches for 12 weeks, to receive either one or four 15-20-minute counseling sessions, and to receive counseling that is either dual focused or smoking focused. Dual Focused Cessation will focus on quitting both smoking and vaping on the target quit date (TQD). Pre-TQD, participants will be instructed to change smoking and vaping patterns (e.g., not smoking or vaping in specific places or at specific times of day). Post-TQD, participants will focus on building smoking and vaping cessation skills (e.g., coping with cravings to smoke or vape, avoiding smoking and vaping cues). Smoking Focused Cessation will focus on quitting smoking on the TQD and using ENDS as a behavioral substitute (i.e., using ENDS as a cigarette substitute). Pre-TQD, participants will be instructed to change smoking patterns (e.g., vaping rather than smoking in specific places or at specific times of day, vaping first in the morning rather than smoking) and practice smoking cessation coping strategies (e.g., substituting ENDS for cigarettes, avoiding smoking cues). Participants will be advised to quit smoking on the TQD and not worry about quitting vaping at this point. Participants will complete daily measures of smoking, vaping, and potential change mechanisms (e.g., craving, smoking reward, self-efficacy) via ecological momentary assessment (EMA) for 2 weeks pre-TQD and 2 weeks post-TQD. Follow-up will occur for 12 months post-TQD.

Primary Objective: Determine which pharmacologic and counseling approaches are especially effective, alone or in combination, in helping dual users quit smoking.

Secondary Objectives:

* Examine the effects of the treatments on variables that may mediate treatment effects on smoking cessation.
* Examine

  1. changes in vaping intensity and vaping cessation
  2. moderators of treatment effects (e.g., cigarette dependence, race, menthol use, ENDS characteristics), and
  3. whether continued vaping is related to cigarette lapse and relapse amongst those who have quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and communicate in English
* Willing to set a quit date to quit smoking cigarettes in the next 30 days
* Willing and medically able to use varenicline and nicotine patches
* Smoking ≥ 5 cigarettes per day for the past 6 months
* Vaping weekly for at least 6 months
* Willing to stop using nicotine replacement or varenicline
* Willing to stop using bupropion (i.e., Wellbutrin, Zyban) if they are currently using it only for smoking cessation
* Saliva cotinine >20 ng/ml
* US resident
* Own a Smartphone to use and download an app to record data

Exclusion Criteria:

* Currently in treatment for psychosis or bipolar disorder
* If they are currently taking bupropion for non-smoking cessation reasons (e.g., Wellbutrin for depression)
* Currently pregnant or breastfeeding. If a participant becomes pregnant while in the study, they will be allowed to continue in the study but will no longer receive study medications. They will also be asked to return any unused study medications.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
52-week biochemically confirmed 7-day point-prevalence abstinence from cigarettes | up to 52 weeks
  52-week biochemically confirmed (anabasine<2 ng/ml) 7-day point-prevalence abstinence from cigarettes

SECONDARY OUTCOMES:
26-week biochemically confirmed 7-day point-prevalence abstinence from cigarettes | up to 26 weeks
  26-week biochemically confirmed (anabasine<2 ng/ml) 7-day point-prevalence abstinence from cigarettes
7-day point-prevalence abstinence from smoking and vaping at Weeks 26 and 52 post-TQD | up to 52 weeks
  Biochemically confirmed with saliva cotinine <30 ng/mL

OTHER OUTCOMES:
Number of Participants Achieving Initial Smoking Abstinence | up to 2 weeks
  Measured by self-reported 24-hours of cigarette abstinence within the first 2 weeks of the target quit day
12-week biochemically confirmed 7-day point-prevalence abstinence from cigarettes | up to 12 Weeks (end of treatment)
  12-week biochemically confirmed (anabasine<2 ng/ml) 7-day point-prevalence abstinence from cigarettes
7-day point-prevalence abstinence from smoking and vaping at Week 12 | up to 12 Weeks (end of treatment)
  Biochemically confirmed with saliva cotinine <30 ng/mL
Number of Participants Achieving Initial Abstinence from Smoking and Vaping | up to 2 weeks
  Measured by self-reported 24-hours of cigarette and ENDS abstinence within the first 2 weeks of the target quit day
Number of days until first cigarette following initial cessation | up to 52 weeks post-TQD
  Latency to lapse (number of days until first cigarette following initial cessation) computed over the full 52 weeks post-TQD
Number of days until 7 consecutive days of smoking following initial cessation | up to 52 weeks post-TQD
  Latency to relapse (number of days until 7 consecutive days of smoking following initial cessation) computed over the full 52 weeks post-TQD.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piper, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF